CLINICAL TRIAL: NCT00468156
Title: Implementation Intentions for Improving Fruit and Vegetable Intakes
Brief Title: The Fruit and Vegetable Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Zora Djuric, Research Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00004225
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2008-11

CONDITIONS: Cancer
Keywords: fruit; vegetables; prevention; cancer; counseling; cancer risk
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): written materials only
  Interventions: Behavioral: written materials only
- 2 (Experimental): written materials plus asked to form implementation intentions
  Interventions: Behavioral: written materials
- 3 (Experimental): same as arm 2 plus telephone support
  Interventions: Behavioral: telephone support

INTERVENTIONS:
Behavioral: written materials only — related to fruit/vegetable servings/day
  Other Names: control
  Arms: 1
Behavioral: written materials — related to fruit/vegetable servings/day
  Other Names: asked to form implementation intentions
  Arms: 2
Behavioral: telephone support — related to fruit/vegetable servings/day
  Other Names: written plus telephone
  Arms: 3

SUMMARY:
The main aim of this study is to determine if persons can increase fruit and vegetable intakes if they make a specific plan to do so.

DETAILED DESCRIPTION:
The conduct of cancer prevention trials through community settings and/or national networks of clinical sites requires the development of appropriate interventions. One promising behavioral strategy that is very simple to administer is that of the formulation of implementation intentions. The premise of this intervention is that once persons formulate a plan of action, automatic behavior follows. Use of this intervention in primary care is an innovative approach to eliciting preventive behaviors with minimal staff time. The goal in this study will be to increase fruit and vegetable consumption by 2 servings/day without a change in overall energy intakes by decreasing consumption of a less nutritious food. Substitution of foods is critical for prevention of weight gain. This feasibility study aims conduct a randomized, controlled clinical trial to test whether formulation of implementation intentions, either alone or with telephone support, can increase fruit and vegetable consumption without an increase in overall energy intakes. Recruitment success in a family medicine clinic in Ypsilanti Michigan will be documented with emphasis on the extent of minority participation. Dietary assessment will be the main outcome variable. Other assessments will include demographics, self-assessment of behaviors targeted by the intervention and levels of carotenoids in plasma. We will enroll 105 subjects to retain 28/arm, and power is good to detect small differences in fruit and vegetable intakes among the three study arms. This will generate useful data for the design of larger dietary intervention trials that are cost-effective and which will utilize multiple clinical sites to optimize enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 and older
* Give informed consent
* In general good health
* Less than 5.5 servings/day of fruits and vegetables

Exclusion Criteria:

* On medically prescribed diets that the study would not be consistent with
* Evidence of eating disorders
* Health problems that affect energy needs (eg. broken leg can interfere with normal activities and affect energy needs).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Document enrollment success at a primary care clinic | 8 months

SECONDARY OUTCOMES:
Determine change in fruit and vegetable consumption | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, PhD, Principal Investigator — University of Michigan
Locations (1):
- Ypsilanti Family Health Center, Ypsilanti, Michigan, United States

REFERENCES:
- [Result] Djuric Z, Ellsworth JS, Ren J, Sen A, Ruffin MT 4th. A randomized feasibility trial of brief telephone counseling to increase fruit and vegetable intakes. Prev Med. 2010 May-Jun;50(5-6):265-71. doi: 10.1016/j.ypmed.2010.03.003. Epub 2010 Mar 11. PMID 20226809